CLINICAL TRIAL: NCT02385864
Title: Effect of the Continuous Positive Airway Pressure on Blood Pressure and Arterial Stiffness in Obstructive Sleep Apnea Patients With Resistant Hypertension
Brief Title: CPAP Effect on Blood Pressure and Arterial Stiffness in Obstructive Sleep Apnea Patients With Resistant Hypertension
Acronym: POP-ART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A00908-37
Record Dates: First submitted 2015-02-26; First posted 2015-03-11 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Hypertension, Resistant to Conventional Therapy; Obstructive Sleep Apnea
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Resistant hypertension is defined as uncontrolled blood pressure (BP ≥ 140/90mmHg) despite the current use of three or more antihypertensive drugs at full doses, including a diuretic. Obstructive Sleep Apnea (OSA) is at high risk for cardiovascular morbidity and is highly prevalent in patients with resistant hypertension.

The prospective observational POP-ART study will assess the efficacy of continuous positive airway pressure (CPAP) treatment on BP in patients with resistant hypertension and collect data from usual care.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea is highly prevalent in patients with resistant hypertension and several studies have assessed the effect of CPAP treatment on BP.

But only few studies have raised data about the effect of CPAP treatment on BP in patients with resistant hypertension.

Hypertension is moreover associated with increased arterial stiffness, but no data are available in patients with resistant hypertension.

The purpose of this study is to demonstrate that OSA has a major impact in resistant hypertension, whose effects on BP and arterial stiffness can partially be reversible with CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with resistant hypertension uncontrolled by 3 or more antihypertensive agents
* Patient with severe OSA (apnea-hypopnea index > 30 or > or equal to 15 with excessive daytime sleepiness), or with mild to moderate OSA without excessive daytime sleepiness, or without OSA.
* Ambulatory patient

Exclusion Criteria:

* Body mass index ≥40 kg/m2
* Other identifiable causes of hypertension
* Contraindication to CPAP treatment or patient already treated with CPAP

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resistant hypertension
Sampling Method: Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-08 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Mean variation in BP at 6 months, assessed by 24h ambulatory BP monitoring | 6 months from baseline assessment

SECONDARY OUTCOMES:
OSA prevalence in patients with resistant hypertension | 6 months
BP variability assessed by home self BP measurments | 6 months
Arterial stiffness assessed by pulse wave velocity and QKD interval | 6 months
Antihypertensive treatment consumption | 6 months
CPAP treatment observance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Baguet, MD, PhD, Principal Investigator — Groupe Hospitalier Mutualiste, Grenoble
Locations (4):
- France (4):
  - Clinique du Tondu, Bordeaux
  - Bordeaux University Hospital, Bordeaux
  - Clinique des Eaux Claires, Groupe Hospitalier Mutualiste, Grenoble
  - Grenoble University Hospital, Grenoble